CLINICAL TRIAL: NCT01802606
Title: Department of Pharmacy, Xijing Hospital
Brief Title: Factors Related to Infection Prevention After Tension-free Inguinal Hernia Repair
Acronym: infection
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20091217
Record Dates: First submitted 2012-10-31; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: INFECTION
Keywords: surgery; administration; infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators conducted the study in 4 teaching hospitals and 2 non-teaching hospitals of Shaanxi Province. Surgeons, clinical pharmacists and nurses took part in patient collection, information registration, protocol performance.

The investigators recruited 1200 patients with inguinal hernia undergoing inguinal hernioplasty in the six hospitals from January 2010 to July 2011. The patients were randomly allocated into control group, cefazolin group and levofloxacin group, with digital meter method , 400 in each group. The data such as age, sex, case number, length of hospital stay, antibiotic usage, post-operative infection, infection site, bacterial culture were filled in self-designed forms on computer.

DETAILED DESCRIPTION:
All of the patients received tension-free inguinal hernia repair with a mesh plug. The surgical-site infection (SSI) was diagnosed according to the criteria of the Centers for Disease Control and Prevention [5-6].

We chose cefazolin sodium and levofloxacin sodium chloride injection as peri-operative antibiotics. Cefazolin sodium is an effective antibiotic with a short plasma elimination half-life against gram-positive cocci (GPC) except for enterococci and meticillin-resistant staphylococci. It is recommended as one of the prior antibacterial agents used for clearing cuts and preventing infection in many countries including China. Levofloxacin sodium chloride injection has a wide anti-bacterial spectrum composed of gram-negative bacteria and gram-positive anaerobic bacteria including anaerobic bacteria. It can remain a high concentration in urine, so it is recommended as an attractive antibiotic for urinary tract operation [5].

In the control group, we gave normal saline as placebo by intravenous drip infusion for 30-60 min before operation. Cefazolin group and levofloxacin group received intravenous administration of cefazolin sodium 1000 mg and levofloxacin sodium chloride injection 200 mg, respectively, for 30-60 min before operation.

ELIGIBILITY:
Inclusion Criteria:

1. males or females aged 16-18 years old;
2. no infection or hematological system disease before surgery;
3. normal liver and kidney function;
4. no pre-operative valvular heart disease;
5. Body mass index (BMI) within 18-32.

Exclusion Criteria:

1. fail to meet one of the inclusion criteria above;
2. malignant tumor;
3. history of immune system diseases;
4. using or had used corticosteroids or immunosuppressants less than 1 month before surgery;
5. using or had used antibiotics less than 3 d before surgery;
6. pregnancy or lactation.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: e recruited 1200 patients with inguinal hernia undergoing inguinal hernioplasty in the six hospitals
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Factors related to infection prevention after tension-free inguinal hernia repair | up to 5 weeks

SECONDARY OUTCOMES:
to offer some evidence pertaining to the factors influencing the prevention of infection and complications after tension-free inguinal hernia repair. | up to 6 months
  Our study aims to offer some evidence pertaining to the factors influencing the prevention of infection and complications after tension-free inguinal hernia repair.

CONTACTS AND LOCATIONS:
Overall Officials: Aidong Wen, pro., Principal Investigator — Xijing Hospital